CLINICAL TRIAL: NCT01381432
Title: Special Drug Use Investigation for IMURAN (Azathioprine) Tablet (Pulmones Transplantation)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112314
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Liver Diseases
Keywords: Antirejection
MeSH Terms: conditions — Liver Diseases | interventions — Azathioprine

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed azathioprine tablet: Subjects prescribed azathioprine tablet during study period after the lung transplantation
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: Azathioprine — At the start of treatment, 2 to 3 mg per kg of body weight each day. For the rest of treatment, 1 to 2 mg per kg of body weight each day.

SUMMARY:
This post-marketing surveillance study is to investigate the efficacy and safety of azathioprine tablets in subjects whom lung transplantation is performed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who undergo lung transplantation and azathioprine tablets were administered

Exclusion Criteria:

* Subjects with hypersensitivity to the ingredients of azathioprine tablet
* Subjects who is pregnant or might be pregnant
* Subjects whose white count is lower than 3000/cubic millimeter

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The following subjects to whom azathioprine tablet is administered for "the suppression of lung transplant rejection";
  1. Subjects on whom lung transplantation is performed after approval and to whom azathioprine tablet is administered from transplant surgery to May 2010.
  2. Subjects on whom lung transplantation is performed before approval and who have already completed the drug administeration as well as during the drug administration at the time of the contract terminiation.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2004-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events related to azathioprine tablets | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline